CLINICAL TRIAL: NCT02561793
Title: Does DHEA Improve Pregnancy Rate in Women Undergoing IVF/Intracytoplasmatic Sperm Injection(ICSI) With Expected Poor Ovarian Response According to the Bologna Criteria? A Double Blind Randomized Placebo Controlled Study
Brief Title: DHEA Versus Placebo in Women With Poor Ovarian Response
Acronym: DHEA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, AbdelGany Hassan, Lecturer of Gynecology and Obstetrics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DHEA 2
Record Dates: First submitted 2015-09-25; First posted 2015-09-28 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Subfertility
MeSH Terms: conditions — Infertility | interventions — Dehydroepiandrosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DHEA (Active Comparator): Women will receive DHEA 12 weeks before starting IVF/ICSI
  Interventions: Drug: DHEA
- Placebo (Placebo Comparator): Women will receive a placebo 12 weeks before starting IVF/ICSI
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DHEA — Women will receive DHEA 12 weeks before starting IVF/ICSI
  Arms: DHEA
Drug: Placebo — women will receive a placebo 12 weeks before starting IVF/ICSI
  Arms: Placebo

SUMMARY:
440 women with expected poor ovarian response undergoing IVF/ICSI (intracytoplasmic sperm injection) will be randomly divided into 2 groups using computer generated random numbers . Group 1 ( study group) will receive Dehydroepiandrosterone (DHEA) 25 mg ( DHEA 25mg, Natrol , USA) t.d.s daily for 12 weeks before starting IVF/ICSI cycle. Group 2 ( control group) will receive a placebo. Patients included in the study will be subjected to full history taking and clinical examination. On the second day of menstruation serum FSH, LH, Prolactin and Oestradiol will be assessed and the antral follicular count (AFC) will be assessed using a vaginal ultrasound scan. AFC will be defined as the number of follicles measuring 3-10mm.

All patients will have gonadotropin antagonist protocol with Human menopausal gonadotrophin (HMG) stimulation until the day of (Human chorionic gonadotrophin (HCG) administration. On the day of HCG administration, ovarian ultrasound scan will be performed using a transvaginal probe. Oocytes will be aspirated 34-36 hours after HCG administration. Oocytes will be fertilized and embryos will be transferred. Both groups will be compared regarding the proportion of pregnancy.

DETAILED DESCRIPTION:
The study will be conducted in Cairo university hospitals and Dar Al-Teb Infertility and Assisted conception center, Giza Egypt. All patients attending the centre will be evaluated for their expected ovarian response.Patients fulfilling the Bologna criteria definition of poor ovarian response will be invited to participate in the study and to sign informed consent forms. The invitation will include a clear full explanation of the study.

440 women will be randomly divided into 2 groups using computer generated random numbers. Group 1 ( study group) will include 220 women who will receive DHEA 25 mg t.d.s ( DHEA®, Natrol , USA) twice daily for 12 weeks before starting IVF/ICSI cycle. Group 2 will include 220 women who will receive an oral placebo similar in colour, size and structure to DHEA.. All women fulfilling the inclusion criteria will be invited to participate in the study. A written informed consent will be taken and only women signing the consent will be included in the study.

Patients included in the study will be subjected to full history taking and clinical examination including general, abdominal and gynecological examination. This will be followed by a vaginal ultrasound scan to assess uterus, ovaries and any pelvic masses.

On the second day of menstruation serum follicle stimulating hormone (FSH), luteinizing hormone (LH) , Prolactin and Oestradiol will be assessed and the antral follicular count (AFC) will be assessed using a vaginal ultrasound scan. AFC will be defined as the number of follicles measuring 3-10mm.

The stimulation protocol will start on day 2 using 450-300 IU HMG ( Merional® IBSA, Lugano, Switzerland) and gonadotropin-releasing hormone antagonist, cetrorelix (Cetrotide® Merck Serono, Darmstadt, Germany) 0.025 mg daily. Gonadotropins will be administered for 4 to 5 days, after which the dose will be adjusted according to the ovarian response. The ovarian response will be monitored by transvaginal ultrasound and serum E2 levels. When three or more follicles reached a maximum diameter of 16 mm, highly purified HCG 5000 or 10,000 IU (Choriomon ®IBSA) will be administered. The procedure will be cancelled if less than 3 follicles 16 mm in size are present 12 days after starting gonadotropins despite doses reaching 450 IU. The cycle will be also cancelled if there is risk of ovarian hyperstimulation like massive ovarian enlargement or serum estradiol exceeds 3000pg/L Transvaginal oocyte retrieval will be performed 34-36 h after the administration of HCG. Oocytes will be fertilized either via IVF or ICSI based on the couple's history. Fertilization will be assessed 16-18 h after IVF or ICSI . Embryos will be transferred on Day 3 or 5. Vaginal tablets containing progesterone (Prontogest® IBSA) 400 mg/day will be given when fertilization is confirmed. A pregnancy test will be done 2 weeks after embryo transfer. For patients with a positive pregnancy test, progesterone is to be continued for an additional 4 weeks. Clinical pregnancy will be defined as Visualization of an intrauterine gestational sac 5 weeks after embryo transfer.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing IVF/ICSI treatment with expected poor ovarian response according to the Bologna criteria

Exclusion Criteria:

* Women with BMI >35 Kg/m2
* Women with a single ovary
* Known allergy to DHEA
* Diabetic women on insulin as insulin lowers DHEA levels and might reduce the effectiveness of DHEA supplements

Ages: 20 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 440 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | 12 weeks after embryo transfer
  Ongoing pregnancy will be confirmed by a transvaginal scan confirming the presence of an embryo with evidence of heart beats.

SECONDARY OUTCOMES:
Clinical pregnancy rate | 5 weeks after embryo transfer
  clinical pregnancy will be confirmed by detecting a gestational sac using a transvaginal ultrasound

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Cairo University Hospitals, Cairo
  - Dar AlTeb subfertility centre, Giza

REFERENCES:
- [Background] Jirge PR, Chougule SM, Gavali VG, Bhomkar DA. Impact of dehydroepiandrosterone on clinical outcome in poor responders: A pilot study in women undergoing in vitro fertilization, using bologna criteria. J Hum Reprod Sci. 2014 Jul;7(3):175-80. doi: 10.4103/0974-1208.142477. PMID 25395742
- [Background] Xu B, Li Z, Yue J, Jin L, Li Y, Ai J, Zhang H, Zhu G. Effect of dehydroepiandrosterone administration in patients with poor ovarian response according to the Bologna criteria. PLoS One. 2014 Jun 16;9(6):e99858. doi: 10.1371/journal.pone.0099858. eCollection 2014. PMID 24932478
- [Background] Spremovic-Radjenovic S, Bila J, Gudovic A, Vidakovic S, Dokic M, Radunovic N. [Poor Ovarian Response to Stimulation for In Vitro Fertilization]. Srp Arh Celok Lek. 2015 May-Jun;143(5-6):354-61. doi: 10.2298/sarh1506354s. Serbian. PMID 26259413